CLINICAL TRIAL: NCT02183870
Title: EUCROSS: A Phase II Trial to Evaluate Efficacy and Safety of Crizotinib Treatment in Advanced Adenocarcinoma of the Lung Harbouring ROS1 Translocations
Brief Title: EUCROSS: European Trial on Crizotinib in ROS1 Translocated Lung Cancer
Acronym: EUCROSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Spanish Lung Cancer Group (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Juergen Wolf, Professor Dr. med., Leader of the LCGC, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUCROSS; 2013-002737-38 (EudraCT Number); DRKS00005409 (Other: DRKS)
Record Dates: First submitted 2014-06-25; First posted 2014-07-08 (Estimated); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Lung Cancer; Adenocarcinoma; NSCLC
Keywords: lung cancer; adenocarcinoma; NSCLC; ROS1; ROS1 translocation; crizotinib; phase II
MeSH Terms: conditions — Lung Neoplasms; Adenocarcinoma | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Crizotinib (Experimental): Patients are treated in this single-arm trial with oral crizotinib 250 mg b.i.d.. Treatment dose will be adjusted according to the protocol if indicated. Treatment will be conducted until disease progression or beyond disease progression according to the protocol if clinically indicated.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Crizotinib — 250mg crizotinib bid until end of treatment
  Other Names: Xalkori

SUMMARY:
EUCROSS is a phase II trial to evaluate the efficacy and safety of crizotinib in patients with adenocarcinoma of the lung harbouring ROS1 translocations. Patients will be treated with 250mg crizotinib bid until progression or intolerable toxicity.

DETAILED DESCRIPTION:
EUCROSS is a phase II trial to evaluate the efficacy and safety of crizotinib in patients with adenocarcinoma of the lung harbouring ROS1 translocations. In individual treatment attempts and an ongoing phase I trial crizotinib has shown remarkable effects on this selected subgroup of lung cancer patients. Crizotinib is a tyrosine kinase inhibitor, blocking the catalytic activity of rearranged ALK and ROS1 as well as MET. The patients eligible for the trial will be treated with 250mg crizotinib twice-daily. Tumor response to treatment will be assessed every 6 weeks by CT or MRI scans. In case of progression treatment beyond may be conducted if clinically indicated. To identify mechanisms of resistance to crizotinib treatment, an optional re-biopsy may be performed in these cases and fresh frozen tumor material will analyzed at the University of Cologne.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adenocarcinoma of the lung that is locally advanced or metastatic independent from the number of prior lines of therapy, i.e. including non-pretreated patients (UICC stage IIIB or IV)
* Positive for ROS1 translocation by central FISH-testing
* Ability to swallow pills
* Age > 18 years
* ECOG performance status 0 to 2
* Life expectancy of at least 12 weeks
* Disease measurable per Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1)
* Any prior treatment (chemotherapy, radiation or surgery) must have been completed at least 2 weeks prior to initiation of study medication
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 14 days prior to screening:
* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count (ANC) ≥ 1,000 /mm3
* Platelet count ≥ 50 000/µL
* Total bilirubin ≤ 2 x upper limit of normal (ULN)
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (AP) ≤ 2,5 x ULN or ≤ 5 x ULN in case of liver involvement
* PT-INR/PTT ≤ 1.5 x ULN
* Serum creatinine ≤ 2 times ULN
* Calculated creatinine clearance (CLcr) ≥ 40 ml/min (Cockcroft-Gault formula)
* Written informed consent
* Negative serum pregnancy test within 3 days prior to start of dosing premenopausal women. Women of non-childbearing potential may be included without serum pregnancy test if they are either surgically sterile or have been postmenopausal for ≥ 1 year.

Fertile men and women must have an effective method of contraception during treatment and for at least 3 months after completion of treatment as directed by their physician. Effective methods of contraception result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly (for example implants, injectables, combined oral contraception or intra-uterine devices). At the discretion of the investigator, acceptable methods of contraception may include total abstinence where lifestyle of the patient ensures compliance (Periodic abstinence and withdrawal are not acceptable methods of contraception).

Exclusion Criteria:

* Previous treatment with specific ALK or ROS1 inhibitors
* Current treatment within another therapeutic clinical trial
* Other history of ongoing malignancy that would potentially interfere with the interpretation of efficacy (early stage or chronic disease is allowed if not requiring active therapy or intervention and being under control)
* Pregnancy or breastfeeding
* Use of drugs or foods that are known potent CYP3A4 inhibitors, including but not limited to atazanavir, clarithromycin, indinavir, itraconazole, ketoconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin, voriconazole and grapefruit or grapefruit juice
* Use of drugs that are known potent CYP3A4 inducers, including but not limited to carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, and St. John's wort
* Use of drugs that are CYP3A4 substrates with narrow therapeutic indices, including but not limited to dihydroergotamine, ergotamine, pimozide, astemizole, cisapride, and terfenadine
* Active CNS metastases. Patients with brain metastasis are eligible if asymptomatic for ≥ 14 days before starting study medication and off corticosteroids.
* History of or known carcinomatous meningitis or leptomeningeal disease
* Known diagnosis of HIV, active hepatitis B and/or C (testing is not mandatory)
* Any person being in an institution on assignment of the respective authority against his/her own will
* Any medical, mental or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or understand the patient information
* Ongoing cardiac dysrhythmias of CTCAE grade ≥2, uncontrolled atrial fibrillation of any grade or QTcF interval > 470ms
* Patients with known interstitial fibrosis or interstitial lung disease
* Any of the following within 3 months prior to first crizotinib administration:

Myocardial infarction, severe/unstable angina, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-05; Primary Completion 2018-07-24 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR); evaluation criteria: investigator assessed RECIST v.1.1 analysis | From time of beginning of treatment until the documention of response according to RECIST v1.1 (expected average 12 months) .
  CT/MRI scans will be performed to evaluate the efficacy of crizotinib treatment in advanced adenocarcinoma of the lung harbouring ROS1 fusion genes (primary outcome measure: objective response rate (ORR) according to RECIST v.1.1)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) according to RECIST v1.1; evaluation criteria: investigator assessed RECIST v.1.1 analysis | From time of beginning of treatment until the first documented event of progression according to RECIST v1.1 (expected average 12 months).
  CT/MRI scans will be performed to assess the PFS during treatment period.
Overall Survival (OS); evaluation criteria: investigator assessed RECIST v.1.1 analysis | From beginning to end of study (Last subject last visit (LSLV)) (up to approximately 24 months).
  OS will be assessed by telephone calls every 3 months after the safety follow-up visit.
Duration of Response (DR); evaluation criteria: investigator assessed RECIST v.1.1 analysis | From time of beginning of treatment until the documention of progression according to RECIST v1.1 (expected average 12 months).
  CT/MRI scans will be performed to asses the DR.
Time to Tumor Response; evaluation criteria: investigator assessed RECIST v.1.1 analysis | From time of beginning of treatment until the first documented event of response according to RECIST v1.1 (expected average 3 months).
  CT/MRI scans will be performed to assess the Time to Tumor Response.
Disease Control Rate (DCR); evaluation criteria: investigator assessed RECIST v.1.1 analysis | From beginning of treatment to week 6, 12 and 24 according to RECIST v1.1 (expected average 3 months).
  CT/MRI scans will be performed at weeks 6, 12, 24 to assess the DCR.
Safety/Adverse Events and tolerability in all patients treated with crizotinib assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram and RECIST1.1 | From beginning of treatment until 28 days post treatment (expected average 12 months).
  Safety and tolerability will be assessed on every study visit and for 28 days after end of treatment.
Patient Reported Outcomes (PRO) (EORTC QLQ-C30, EORTC QLQ-LC13) | Questionnaires (EORTC QLQ-LC13, EORTC QLQ-C30) completed at baseline and every 4 weeks from beginning of treatment until end of study.
  Patient reported outcomes (PRO) of health-related quality of life (HRQoL), disease/treatment related symptoms of lung cancer and general health status
To evaluate the efficacy of crizotinib treatment in the patient subgroup with ROS1 translocation confirmed by the CAGE technology regarding the objective response rate (ORR) (evaluation criteria: investigator assessed RECIST v1.1) | From time of beginning of treatment until the documention of response according to RECIST v1.1 (expected average 12 months) .
  CT/MRI scans will be performed to evaluate the efficacy of crizotinib treatment in advanced adenocarcinoma of the lung harbouring ROS1 fusion genes as confirmed by CAGE sequencing
Objective Response Rate (ORR), Overall Survival (OS), Progression Free Survival (PFS), Duration of Response (DR), Time to Tumor Response, Disease Control Rate (DCR); evaluation criteria: RECIST v1.1 by independent radiologic review | From time of beginning of treatment until the documention of response according to RECIST v1.1 (expected average 12 months) .
  CT/MRI scans will be performed to evaluate the efficacy of crizotinib treatment

OTHER OUTCOMES:
Characterization of ROS1 fusion gene on a genomic level by CAGE Technology to identify the exact break-apart point as well as the involved fusion genes. | From beginning of screening of first patient to screening of last patient (expected average 24 months).
  CAGE technology (Cap Analysis of Gene Expression) is an RNA based sequencing technology to identify the exact break-apart point as well as the fusion genes.
Characterization of molecular and genetic mechanisms of resistance to crizotinib treatment in patients showing disease progression. | At time of disease progression (expected average 12 months).
  Mechanisms of resistance to crizotinib will be analysed by molecular pathologic analyses, e.g. NGS and FISH.

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Wolf, Prof. Dr. med., Principal Investigator — Uniklinik Köln, Department I for Internal Medicine, LCGC
Locations (18):
- Germany (6):
  - Thoraxklinik Heidelberg, Heidelberg, Baden-Würtemberg
  - Universitätsklinikum Frankfurt - Medizinische Klinik II, Frankfurt a.M., Hesse
  - LungenClinic Großhansdorf, Großhansdorf, Schleswig-Holstein
  - Evangelische Lungenklinik Berlin, Berlin
  - University of Cologne / LCGC, Cologne
  - Universitätsklinikum Tübingen, Tübingen
- Spain (11):
  - Maria Rosaria Garcia Campelo, A Coruña
  - CEIC Hospital General Universitario de Alicante, Alicante
  - CEIC Hopsital Vall d'Hebron, Barcelona
  - Institut Catala D'Oncologia, Barcelona
  - Hospital Universitario Materno-Infantil de Canarias, Las Palmas de Gran Canaria
  - CEIC Área 2 - Hospital Universitario de La Princesa, Madrid
  - CEIC Área 6 - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - CEIC Malaga Nordeste - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Son Llatzer, Palma de Mallorca
  - CEIC Hospital Universitario Virgen del Rocio, Seville
  - CEIC Hospital Clínico Universitario de Valencia, Valencia
- Universitätsspital Basel, Basel, Switzerland

REFERENCES:
- [Background] Bos M, Gardizi M, Schildhaus HU, Heukamp LC, Geist T, Kaminsky B, Zander T, Nogova L, Scheffler M, Dietlein M, Kobe C, Holstein A, Maintz D, Buttner R, Wolf J. Complete metabolic response in a patient with repeatedly relapsed non-small cell lung cancer harboring ROS1 gene rearrangement after treatment with crizotinib. Lung Cancer. 2013 Jul;81(1):142-3. doi: 10.1016/j.lungcan.2013.02.018. Epub 2013 Apr 1. PMID 23558310
- [Background] Takeuchi K, Soda M, Togashi Y, Suzuki R, Sakata S, Hatano S, Asaka R, Hamanaka W, Ninomiya H, Uehara H, Lim Choi Y, Satoh Y, Okumura S, Nakagawa K, Mano H, Ishikawa Y. RET, ROS1 and ALK fusions in lung cancer. Nat Med. 2012 Feb 12;18(3):378-81. doi: 10.1038/nm.2658. PMID 22327623